CLINICAL TRIAL: NCT03908567
Title: Multicenter Randomized Controlled Phase 2 Trial to Evaluate AM-125 in the Treatment of Acute Peripheral Vertigo Following Neurosurgery (TRAVERS)
Brief Title: AM-125 in the Treatment of Acute Peripheral Vertigo Following Neurosurgery
Acronym: TRAVERS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-125-CL-18-01; 2018-002474-52 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Vestibular Vertigo
Keywords: Vertigo; Balance
MeSH Terms: conditions — Vertigo | interventions — Administration, Intranasal; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For intranasal subjects, allocation is blinded. The oral arm is an open-label arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Nasal spray solution without active ingredient
  Interventions: Other: Intranasal Placebo
- 1 mg AM-125 (Experimental): Nasal spray solution with 5 mg/mL betahistine dihydrochloride. Administered three times daily as 1 spray per nostril. Total daily dose is 3 mg betahistine dihydrochloride.
  Interventions: Drug: Intranasal Drug
- 10 mg AM-125 (Experimental): Nasal spray solution with 50 mg/mL betahistine dihydrochloride. Administered three times daily as 1 spray per nostril. Total daily dose is 30 mg betahistine dihydrochloride.
  Interventions: Drug: Intranasal Drug
- 20 mg AM-125 (Experimental): Nasal spray solution with 100 mg/mL betahistine dihydrochloride. Administered three times daily as 1 spray per nostril. Total daily dose is 60 mg betahistine dihydrochloride.
  Interventions: Drug: Intranasal Drug
- Oral 16 mg betahistine (Experimental): Tablets containing betahistine dihydrochloride. Administered three times daily as 1 tablet per time. Total daily dose is 48 mg oral betahistine dihydrochloride.
  Interventions: Drug: Oral Tablet

INTERVENTIONS:
Drug: Intranasal Drug — Intranasal administration of solution with betahistine dihydrochloride; Dosing 3 times a day
  Arms: 1 mg AM-125; 10 mg AM-125; 20 mg AM-125
Drug: Oral Tablet — Oral dosing with tablets 3 times a day
  Arms: Oral 16 mg betahistine
Other: Intranasal Placebo — Intranasal administration of solution without betahistine dihydrochloride; Dosing 3 times a day
  Arms: Placebo

SUMMARY:
Treatment of vertigo after removal of a tumor of the balance and hearing nerve after neurosurgery, which damages or cuts the vestibular nerve (balance).

This trial explores the efficacy and safety of AM-125 in the treatment of acute vertigo. In this proof of concept trial patients experiencing vertigo after neurosurgery (vestibular schwannoma labyrinthectomy and vestibular neurectomy) will receive AM-125 or placebo. It evaluates the potential of AM-125 versus placebo in reducing the symptoms of vestibular dysfunction and accelerating vestibular compensation following neurosurgery.

ELIGIBILITY:
Main Inclusion Criteria:

1. Scheduled for neurosurgery (vestibular schwannoma resection, labyrinthectomy or vestibular neurectomy).
2. Small to moderately large vestibular schwannoma (Koos grade I-III; Samii grade T1-T3b; ≤ 30 mm in diameter in cerebellopontine angle) that does not displace the brainstem, documented by magnetic resonance imaging not older than six months or Indication for labyrinthectomy or vestibular neurectomy.
3. Confirmed vestibular function on both sides.

Main Exclusion Criteria:

1. Prior radiotherapy (gammaknife, intensity modulated radiation therapy) irradiating the brain-stem with more than 4 Gy.
2. Any ongoing other peripheral vestibular disorder (e.g. Meniere's disease, benign paroxysmal vertigo, vestibular neuritis) or central vestibular disorder (e.g. vestibular migraine, central vertigo).
3. Vestibular rehabilitation therapy or presurgical gentamicin therapy (i.e. "pre-habilitation therapy") within the past three months prior neurosurgery.
4. Any clinically relevant nasal obstruction or pathology precluding effective and/or safe intranasal delivery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Improvement of time standing on foam (eyes closed) | Day 3 to Day 14
Improvement in tandem Romberg test (eyes closed) | Day 3 to Day 14
  Participants will be asked to stand straight in tandem stand (heel of one foot touching the toes of the other foot) and duration in this position will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- CHP Clairval, Marseille, France

REFERENCES:
- See also: Link to Result entry in clinicaltrialsregister.eu — https://www.clinicaltrialsregister.eu/ctr-search/trial/2018-002474-52/results
- See also: Link to peer-reviewed publication of study — https://pubmed.ncbi.nlm.nih.gov/37026797/